CLINICAL TRIAL: NCT00624364
Title: Comparison of Efficacy and Safety of Biphasic Insulin Aspart Plus Metformin to Biphasic Insulin Aspart Monotherapy in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Biphasic Insulin Aspart 30 With Metformin in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1579
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Drug: metformin

SUMMARY:
This trial is conducted in Africa. The aim of this trial is to evaluate the efficacy and safety of biphasic insulin aspart plus OAD compared to biphasic insulin aspart alone on blood glucose control in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with maximum doses of any kind of OAD alone or any kind of oral combination therapy for at least 2 months
* Body mass index (BMI) below 40.0 kg/m2
* HbA1c between 7.5-13.0%

Exclusion Criteria:

* History of drug or alcohol dependence
* Mental incapacity, unwillingness or language barriers precluding adequate
* Subjects previously screened to participation or having already participated in this trial
* Receipt of any investigational drug within the last month prior to this trial
* Known or suspected allergy to trial products or related products

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-05; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 24 weeks of treatment

SECONDARY OUTCOMES:
Plasma glucose profiles
Cardiovascular risk factors
Incidence of hypoglycaemic episodes
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (11):
- South Africa (11):
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Pietermaritzburg, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Benoni
  - Novo Nordisk Investigational Site, Bloemfontein
  - Novo Nordisk Investigational Site, Kimberley
  - Novo Nordisk Investigational Site, Richards Bay

REFERENCES:
- [Result] Naiker P, Makan HA, Kedijang T, Kong LLL, Omar MAK & the BIAsp-1579 Study Group. Effects of Once-Daily Biphasic Insulin Aspart 30 with Metformin versus Twice-Daily Biphasic Insulin Aspart 30 in South African Type 2 Diabetes Subjects. Society for Endocrinology, Metabolism and Diabetes of South Africa (SEMDSA); Country: South Africa City: Bloemfontein
- [Result] Naiker P, Makan HA, Omar MAK, Kedijang T, Kong LLL, the BIAsp-1579 Study Group. Effect of biphasic insulin aspart 30/70 (BIAsp30) in combination with metformin on glycaemic control in subjects with type 2 diabetes not optimally controlled on oral antidiabetic agents. EASD 2006 2006; 49(Suppl 1): 599
- [Result] Naiker P, Makan HA, Omar MAK, Kedijang T, Kong LLL, the BIAsp-1579 Study Group. Efficacy of biphasic insulin aspart 30/70 with metformin on glycaemic control in poorly-controlled type 2 diabetes. IDF 2006 2006; 23(Suppl 4): 339 (P940)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com